CLINICAL TRIAL: NCT02815007
Title: Chidamide With EGFR-TKI for Advanced EGFR-TKI-resistant Non-Small Cell Lung Cancer: An Open-label, Single-armed Phase II Trial
Brief Title: Chidamide With EGFR-TKI for Advanced EGFR-TKI-resistant Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yuankai Shi (Other)
Responsible Party: Sponsor-Investigator, Yuankai Shi, Doctor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CancerIHCAMS
Record Dates: First submitted 2016-06-19; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Advanced EGFR-TKI-resistant Non-Small Cell Lung Cancer
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chidamide with EGFR-TKI (Experimental): Chidamide: Per Os, 30mg (5mg*6), twice a week, time interval between 2 medications should be ≥3 days, medicine taken 30 minutes after breakfast.
  EGFR-TKI:
  Taken according to the instruction book
  Interventions: Drug: Chidamide with EGFR-TKI

INTERVENTIONS:
Drug: Chidamide with EGFR-TKI — Chidamide and EGFR-TKI, dosage described in arm description.
  Other Names: Epidaza，HBI-8000

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Chidamide with EGFR-TKI for Advanced EGFR-TKI-resistant Non-Small Cell Lung Cancer

DETAILED DESCRIPTION:
(1)The efficacy of the regimen is evaluated by objective remission rate, disease control rate, progress free survival, duration of remission, overall survival, time to progression.

Safety is monitored by vital signs, blood routine test, liver function, kidney function and electrolytes level, ECG, and cardiac ultrasonography.

All the data is documented by CRF form, and carefully preserved.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IIIB/IV non-small cell lung carcinoma with EGFR 19/21 point mutation, verified by histology or cytology.
2. Achieved remission (CR or PR) over previous EGFR-TKI treatment; or achieved stable disease (SD) ≥ 6 months over previous EGFR-TKI treatment; disease progression emerged during the following EGFR-TKI treatment (within the past 30 days); no other treatment employed after the withdrawn of EGFR-TKI.
3. Age ≥18 years, male or female;
4. Has at least 1 measurable focus according to RECIST criteria 1.1, which has not been treated by radiotherapy.
5. General condition should be ECOG 0-2, expected survival ≥ 3 months.
6. Organ functions should fit the following:

   Bone marrow: absolute neutrophil count ≥1.5 × 109/L, platelet ≥100 × 109/L, Hb ≥ 90g/L; Liver: Total bilirubin ≤ 1.5 times of the normal maximum, ALT and AST≤ 2.5 times of the normal maximum. (ALT/AST≤ 5 times of the normal maximum for patients with infiltrative liver disease) Coagulation: INR or PT ˂ 1.5 folds of the normal maximum; Serum creatinine ˂ 1.5 folds of the normal maximum; creatinine clearance rate ≥50ml/min (calculated by Cockroft-Gault10 formula), for underweight patients, or whose results differ largely from the two formula, other methods for creatinine clearance rate calculation should be employed, like the EDTA method, inulin clearance method or 24 hour urine analysis.
7. For patients with metastatic brain disease, their symptoms should be well controlled by regional therapy (surgery or radiotherapy), and no need for hormone maintenance therapy.
8. For fertile women, urine or blood pregnancy test should be negative within 7 days prior to the treatment, all patients (male and female) should have contraceptive measures during the whole treatment period and 4 weeks after the treatment; willing to sign the written consent and be enrolled in the trial, and adhere to the treatment and follow up protocol.

Exclusion Criteria:

1. Non-small cell lung carcinoma that has not been treated by EGFR-TKI.
2. Patients that have taken other un-authorized medicine or medicine from other trials within 30 days before the 1st day of this trial.
3. Patients with active hemorrhage or new thrombotic disorders, or those who is taking anti-coagulation drugs or those with hemorrhagic tendencies.
4. History of surgery of visceral organs within 6 weeks before the trial.
5. Patients' organ conditions:

   Metastatic brain/ meningeal disorders (except for those whose symptoms are well controlled by regional therapy, and no need for hormone maintenance therapy).

   Patients with history of mesenchymal lung disease, drug-induced mesenchymal disease, hormone-required radiation pneumonia, idiopathic lung fibrosis in baseline CT scan, uncontrolled massive pleural effusion or pericardial effusion.

   Patients with evidence of severe or uncontrolled systemic disease (like unstable or non-compensated respiratory/cardiac/hepatic/renal disease), according to the judgment of the researchers.

   Any unstable systemic disease (including ˃ CTCAE 2 active clinical infection, level IV hypertension, unstable angina pectoris, congestive heart failure, QT interval ˃450ms, HIV infection, metabolic liver or kidney disease); History of any malignant tumor within 5 years prior to the trial. Definitive history of neural or mental disorders, including seizure or dementia.

   Patients with xenogenic organ transplantation, patients had severe injury or massive surgery 4 weeks prior to the 1st dosage admission of medicine in the trial.
6. Women during pregnancy or lactation.
7. Allergic constitution, like those who are allergic to ≥2 foods or drugs, or allergic to the components of the medicine used in the trial;
8. Any condition that impairs the patients' ability to swallow, and any condition that impairs drug absorption or drug kinetic parameters, including any kind of gastrointestinal resection or surgery;
9. Patients with drug abuse, or any medical, psychological, social conditions that may impair trial process or the evaluation of the results of the trial;
10. Any condition that may influence the safety or compliance of the patients.
11. Patients that the researchers think are not appropriate for regimen in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Objective Remission Rate | through study completion, an average of 15 months
Disease Control Rate | through study completion, an average of 15 months

SECONDARY OUTCOMES:
Progression free survival | through study completion, an average of 15 months
Duration of Remission | through study completion, an average of 15 months
Overall Survival | through study completion, an average of 15 months
Time to Progression | through study completion, an average of 15 months
Vital signs | Every 2 weeks for the first 6 months, every month for the remaining 6 months
Serum alanine aminotransferase level | Every 2 weeks for the first 6 months, every month for the remaining 6 months
Serum aspartate transaminase level | Every 2 weeks for the first 6 months, every month for the remaining 6 months
Serum creatinine level | Every 2 weeks for the first 6 months, every month for the remaining 6 months
Serum urea nitrogen level | Every 2 weeks for the first 6 months, every month for the remaining 6 months
Serum electrolytes level | Every 2 weeks for the first 6 months, every month for the remaining 6 months
Serum brain natriuretic peptide (BNP) level | Every 2 weeks for the first 6 months, every month for the remaining 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Doctor, Principal Investigator — Cancer institute and hospital, Chinese academy of medical sciencees

IPD SHARING:
Plan to Share IPD: Undecided